CLINICAL TRIAL: NCT04250259
Title: A Multi-center, Randomized, Placebo-controlled Trial of S-Adenosylmethionine (SAMe) in Patients With Alcoholic Cirrhosis
Brief Title: SAMe Trial for Patients With Alcoholic Cirrhosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Cedars-Sinai Medical Center (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Suthat Liangpunsakul, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SAMe Trial; 5U01AA026817-04 (NIH)
Record Dates: First submitted 2020-01-22; First posted 2020-01-31 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Alcoholic Cirrhosis
Keywords: Child Class A or B
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic | interventions — S-Adenosylmethionine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Alcoholic Cirrhosis on placebo
  Interventions: Drug: Placebo
- 1,200 mg SAMe (Experimental): SAMe supplement (SAMe 400 mg tablet), 2 tablets in the morning before breakfast and one tablet in the evening before dinner (a total dose of 1,200 mg daily) for 24 months
  Interventions: Drug: SAMe 400 mg tablet
- Non-drinking Controls (No Intervention): Non-drinking healthy controls

INTERVENTIONS:
Drug: Placebo — 2 tablets of placebo in the morning before breakfast and one tablet of placebo in the evening before dinner for 24 months
  Arms: Placebo
Drug: SAMe 400 mg tablet — SAMe supplement (SAMe 400 mg tablet), 2 tablets in the morning before breakfast and one tablet in the evening before dinner (a total dose of 1,200 mg daily) for 24 months
  Arms: 1,200 mg SAMe

SUMMARY:
The proposed of this randomized, double blinded, placebo-controlled study is to assess the effect of SAMe compared to placebo in patients with alcoholic cirrhosis Child Class A and B. The primary objective of the study is to test relationship between SAMe (S-adenosylmethionine) supplement on liver function. The hypothesis is that SAMe supplement will improve liver function in patients with alcoholic liver disease. The improvement in liver function will lead to the reduction in all-cause mortality in patients with alcoholic cirrhosis in those who receive SAMe supplement when compared to those receiving placebo.

ELIGIBILITY:
Inclusion criteria for patients with alcoholic cirrhosis

1. Evidence of cirrhosis as per clinical signs and/or noninvasive transient elastography (Fibroscan®), computed tomography, magnetic resonance imaging including MRI elastography compatible with cirrhosis and/or histopathology by biopsy and
2. subjects with clinical presentation either in Child Class A or B at the time of enrollment
3. individuals 18 to 70 years old and may or may not consume alcohol during study.

Inclusion criteria for healthy control :

) individuals 18 to 70 years old (2) able to provide informed consent (3) subjects do not consume any alcohol or those who drink < 50 grams per day on average in women and < 80 grams per day on average in men (4) subjects are healthy without underlying acute or chronic medical conditions.

Exclusion criteria for patients with alcoholic cirrhosis

1. Active infection as evidenced by positive urine culture, blood culture, or pneumonia,
2. Known co-existing infection with hepatitis C, hepatitis B, or HIV
3. Significant systemic or major illness including chronic obstructive pulmonary disease, congestive heart failure, and renal failure that in the opinion of the Investigator would preclude the patient from participating in and completing the study
4. Gastrointestinal bleeding within the prior 28 days3
5. Participation in another investigational drug, biologic, or medical device trial within 30 days prior to screening
6. Women who are pregnant, may become pregnant, or nursing
7. Presence of any other disease or condition that is interfering with the absorption, distribution, metabolism, or excretion of SAMe such as those with gastric bypass surgery
8. Subjects with history of/diagnosis of hepatocellular carcinoma
9. Members from the same family of study participant. This is based on the recent paper on the non-random sampling in randomized controlled trials4. We acknowledge that if we assign family members to identical treatment, randomization would not be totally correct; but if properly randomized, there is a chance that the members of the family might mix the pills. To avoid this issue and maintain the integrity of randomized blinded fashion, we will not include members from the same family into the study
10. Subjects with psychiatric illnesses such as bipolar disorders as SAMe may interfere with the levels of anti-psychotic drugs and
11. Subjects who are immunocompromised

Exclusion criteria for all healthy control participants:

1. subjects with an active and serious medical disease
2. subjects with an infectious disease
3. consume any alcohol within 3 months before the study
4. subjects with localized or systemic infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
SAMe supplement's effect on all-cause mortality | Baseline to end of 24 months
  The hypothesis is that SAMe supplement will improve liver function in patients with alcoholic liver disease. The improvement in liver function will lead to the reduction in all-cause mortality in patients with alcoholic cirrhosis in those who receive SAMe supplement when compared to those receiving placebo.

SECONDARY OUTCOMES:
SAMe supplement's effect on intestinal permeability function, as defined by serum lipopolysaccharides (LPS) | baseline to end of 24 months
  The function of intestinal permeability will be evaluated by testing serum lipopolysaccharides (LPS) in patients who receive SAMe compared to those who receive placebo. Lipopolysaccharides (LPS) are large molecules consisting of a lipid and a polysaccharide that are bacterial toxins.
SAMe supplement's effect on cellular oxidative stress and/or endoplasmic reticulum (ER) stress, as defined by mitochondrial DNA | baseline to 24 months
  Cellular oxidative stress and/or endoplasmic reticulum (ER) stress will be evaluated by measuring the levels of mitochondrial DNA in the blood of patients who receive SAMe compared to those who receive placebo.
SAMe supplement's effect on liver deuteriation | baseline to 24 months
  determining Proportion of subjects undergoing liver transplantation in patients who receive SAMe compared to those who receive placebo
SAMe supplement's effect on liver developing cancer | baseline to 24 months
  Proportion of subjects developing new onset hepatocellular carcinoma in patients who receive SAMe compared to those who receive placebo
SAMe supplement's effect on infections of the liver | baseline to 24 months
  Proportion of subjects with infection/sepsis (other than SBP) in patients who receive SAMe compared to those who receive placebo
SAMe supplement's effect on other parts of the body | baseline to 24 months
  capture safety-related endpoints by determining proportion of patients with nausea and emesis, proportion of subjects with unexplained diarrhea in patients receive SAMe compared to those who receive placebo.
SAMe supplement's effects on intestinal permeability function, as defined by soluble(s) CD14 | baseline to 24 months
  The function of intestinal permeability will be evaluated by testing soluble(s) CD14 in patients who receive SAMe compared to those who receive placebo. sCD14 either appears after shedding of mCD14 (48 kDa) or is directly secreted from intracellular vesicles (56 kDa).
SAMe supplement's effects on intestinal permeability function, as defined by soluble(s) CD163 | baseline to 24 months
  The function of intestinal permeability will be evaluated by testing soluble(s) CD163 in patients who receive SAMe compared to those who receive placebo. CD163 is an endocytic receptor for haptoglobin-hemoglobin complexes and is expressed solely on macrophages and monocytes. As a result of ectodomain shedding, the extracellular portion of CD163 circulates in blood as a soluble protein (sCD163).
SAMe supplement's effects on cellular oxidative stress and/or endoplasmic reticulum (ER) stress, as defined by cytochrome P450 2E1 levels | baseline to 24 months
  Levels of cellular oxidative stress and/or endoplasmic reticulum (ER) stress will be evaluated by measuring the levels of cytochrome P450 2E1 (CYP2E1) enriched microparticles in patients who receive SAMe compared to those who receive placebo.CYP2E1 is a member of the cytochrome P450 mixed-function oxidase system, which is involved in the metabolism of xenobiotics in the body.

OTHER OUTCOMES:
Exploratory outcome - identify who will improve their liver functions by taking the SAMe supplement amongst those that have been diagnosed with alcoholic cirrhosis (Child-Pugh score of A or B). | baseline to 24 months
  The metabolic profiling of the serum and urine will be collected by those in the study who received the SAMe supplement and will be used as the surrogates for this prediction.

CONTACTS AND LOCATIONS:
Overall Officials: Suthat Liangpunsakul, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Indiana University Hospital, Indianapolis, Indiana